CLINICAL TRIAL: NCT04095988
Title: Allogeneic Microbiota-reconstitution (AMR) for the Treatment of Patients With Diarrhea-predominant Irritable Bowel Syndrome - the AMIRA Trial
Brief Title: Allogeneic Microbiota-reconstitution (AMR) in Diarrhea-predominant Irritable Bowel Syndrome (IBS-D)
Acronym: AMIRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Ulm (Other)
Collaborators: Klinikum Ludwigsburg (Other); Helios Klinikum Krefeld (Unknown); Charite University, Berlin, Germany (Other); Assign International, Berlin, Germany (Unknown)
Responsible Party: Principal Investigator, Thomas Seufferlein, Director Department of Internal Medicine I, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMIRA; 2016-002550-20 (EudraCT Number)
Record Dates: First submitted 2016-06-14; First posted 2019-09-19 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome
Keywords: Allogeneic microbiota reconstitution; diarrhea-predominant irritable bowel syndrome; microbiome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum-AMR (Experimental): Patients receiving Verum-Allogeneic Microbiota Reconstitution via gastroscopy
  Interventions: Procedure: Allogeneic microbiota reconstitution
- Placebo-AMR (Placebo Comparator): Patients receiving Placebo(Saline)-Infusion via gastroscopy
  Interventions: Procedure: Placebo-Allogeneic microbiota reconstitution

INTERVENTIONS:
Procedure: Allogeneic microbiota reconstitution — gastroscopic microbiota Infusion (Verum)
  Arms: Verum-AMR
Procedure: Placebo-Allogeneic microbiota reconstitution — gastroscopic saline Infusion (placebo)
  Arms: Placebo-AMR

SUMMARY:
The investigators will perform a multicenter, 2:1 randomized, double-blinded, placebo-controlled trial of AMR in patients with diarrhea predominant-IBS (IBS-D) diagnosed according to Rome III criteria and the IBS-QOL questionnaire. Central supply and quality control of donor material will be used to control bias.

Primary endpoint is improvement of IBS-SSS (Severity Score System) compared to baseline. Secondary endpoints include changes in IBS-QOL, short term safety and one year follow up to control long term effects, safety and changes in and acceptance of donor microbiome after AMR using16S rDNA sequencing and quantitative diversity analysis.

DETAILED DESCRIPTION:
This study assesses allogeneic microbiota reconstitution (AMR) as novel treatment to improve symptoms and quality of life of patients with diarrhea-predominant irritable bowel syndrome (IBS-D).

The investigators will perform a prospective multicenter, 2:1 randomized, double-blinded, placebo-controlled trial of AMR in patients with IBS-D diagnosed according to Rome III criteria and the IBS-QOL questionnaire.

The experimental intervention is an infusion of donor feces via gastroscopy. The placebo intervention is an infusion of sterile saline via gastroscopy.

Planned number of patients included in the study: 42 patients Planned per-protocol group: 33 patients

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* irritable bowel syndrome of diarrhea-predominant type according to ROME III criteria
* Symptoms for > 1 year before study inclusion
* persisting symptoms > 1 year before study inclusion
* relevant symptoms with reduced Quality of Life (IBS-QOL < 60 Points)
* no specific findings in gastroscopy and colonoscopy with biopsies in the last 2 years

Exclusion Criteria:

* chronic inflammatory diseases
* gastrointestinal infectious diseases
* microscopic colitis
* celiac disease
* diarrhea caused by fructose- or lactose intolerance
* gastrointestinal malignancies or intestinal polyps
* irritable bowel syndrome of other type than IBS-D
* bile acid diarrhea
* constipation
* symptoms caused by other diseases than IBS-D
* dementia
* abdominal surgery in the last months
* antibiotic therapy in the last 3 months
* pregnancy
* linguistic barrier for informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Decrease of the IBS-SSS questionnaire > 105 Points compared to baseline | 90 days after intervention

SECONDARY OUTCOMES:
Improvement of IBS-QOL using IBS-QOL-questionnaire compared to baseline | 90 days and 1 year after intervention
Changes and acceptance of donor microbiome (16S rDNA-analysis) | 90 days after intervention
  16S rDNA-analysis for microbiome biodiversity, correlation to IBS-Symptom Severity Score (IBS-SSS)
Number of participants with treatment related adverse events | follow-up 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas TW Seufferlein, Prof. Dr., Principal Investigator — University Hospital Ulm; Martin Wagner, Prof. Dr., Study Director — University Hospital Ulm; Thomas Frieling, Prof. Dr., Principal Investigator — Helios Klinikum Krefeld
Locations (2):
- Germany (2):
  - Helios Klinikum Krefeld, Krefeld
  - Ulm University Hospital, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borody TJ, George L, Andrews P, Brandl S, Noonan S, Cole P, Hyland L, Morgan A, Maysey J, Moore-Jones D. Bowel-flora alteration: a potential cure for inflammatory bowel disease and irritable bowel syndrome? Med J Aust. 1989 May 15;150(10):604. doi: 10.5694/j.1326-5377.1989.tb136704.x. No abstract available. PMID 2783214
- [Background] Carroll IM, Ringel-Kulka T, Siddle JP, Ringel Y. Alterations in composition and diversity of the intestinal microbiota in patients with diarrhea-predominant irritable bowel syndrome. Neurogastroenterol Motil. 2012 Jun;24(6):521-30, e248. doi: 10.1111/j.1365-2982.2012.01891.x. Epub 2012 Feb 20. PMID 22339879
- [Background] Crouzet L, Gaultier E, Del'Homme C, Cartier C, Delmas E, Dapoigny M, Fioramonti J, Bernalier-Donadille A. The hypersensitivity to colonic distension of IBS patients can be transferred to rats through their fecal microbiota. Neurogastroenterol Motil. 2013 Apr;25(4):e272-82. doi: 10.1111/nmo.12103. Epub 2013 Feb 25. PMID 23433203
- [Background] El-Serag HB, Olden K, Bjorkman D. Health-related quality of life among persons with irritable bowel syndrome: a systematic review. Aliment Pharmacol Ther. 2002 Jun;16(6):1171-85. doi: 10.1046/j.1365-2036.2002.01290.x. PMID 12030961
- [Background] Frieling T, Meis K, Kolck UW, Homann J, Hulsdonk A, Haars U, Hertfelder HJ, Oldenburg J, Seidel H, Molderings GJ. Evidence for mast cell activation in patients with therapy-resistant irritable bowel syndrome. Z Gastroenterol. 2011 Feb;49(2):191-4. doi: 10.1055/s-0029-1245707. Epub 2011 Feb 4. PMID 21298604
- [Background] Grehan MJ, Borody TJ, Leis SM, Campbell J, Mitchell H, Wettstein A. Durable alteration of the colonic microbiota by the administration of donor fecal flora. J Clin Gastroenterol. 2010 Sep;44(8):551-61. doi: 10.1097/MCG.0b013e3181e5d06b. PMID 20716985
- [Background] Hamilton MJ, Weingarden AR, Unno T, Khoruts A, Sadowsky MJ. High-throughput DNA sequence analysis reveals stable engraftment of gut microbiota following transplantation of previously frozen fecal bacteria. Gut Microbes. 2013 Mar-Apr;4(2):125-35. doi: 10.4161/gmic.23571. Epub 2013 Jan 18. PMID 23333862
- [Background] Kajander K, Myllyluoma E, Rajilic-Stojanovic M, Kyronpalo S, Rasmussen M, Jarvenpaa S, Zoetendal EG, de Vos WM, Vapaatalo H, Korpela R. Clinical trial: multispecies probiotic supplementation alleviates the symptoms of irritable bowel syndrome and stabilizes intestinal microbiota. Aliment Pharmacol Ther. 2008 Jan 1;27(1):48-57. doi: 10.1111/j.1365-2036.2007.03542.x. Epub 2007 Oct 5. PMID 17919270
- [Background] Kashyap PC, Marcobal A, Ursell LK, Larauche M, Duboc H, Earle KA, Sonnenburg ED, Ferreyra JA, Higginbottom SK, Million M, Tache Y, Pasricha PJ, Knight R, Farrugia G, Sonnenburg JL. Complex interactions among diet, gastrointestinal transit, and gut microbiota in humanized mice. Gastroenterology. 2013 May;144(5):967-77. doi: 10.1053/j.gastro.2013.01.047. Epub 2013 Feb 1. PMID 23380084
- [Background] Keller J, Wedel T, Seidl H, Kreis ME, Andresen V, Preiss JC, Layer P, van der Voort I. [S3 guideline of the German Society for Digestive and Metabolic Diseases (DGVS) and the German Society for Neurogastroenterology and Motility (DGNM) to the definition, pathophysiology, diagnosis and treatment of intestinal motility]. Z Gastroenterol. 2011 Mar;49(3):374-90. doi: 10.1055/s-0029-1245993. Epub 2011 Mar 9. No abstract available. German. PMID 21391171
- [Background] Longstreth GF, Thompson WG, Chey WD, Houghton LA, Mearin F, Spiller RC. Functional bowel disorders. Gastroenterology. 2006 Apr;130(5):1480-91. doi: 10.1053/j.gastro.2005.11.061. PMID 16678561
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Ohman L, Simren M. Pathogenesis of IBS: role of inflammation, immunity and neuroimmune interactions. Nat Rev Gastroenterol Hepatol. 2010 Mar;7(3):163-73. doi: 10.1038/nrgastro.2010.4. Epub 2010 Jan 26. PMID 20101257
- [Background] Parkes GC, Rayment NB, Hudspith BN, Petrovska L, Lomer MC, Brostoff J, Whelan K, Sanderson JD. Distinct microbial populations exist in the mucosa-associated microbiota of sub-groups of irritable bowel syndrome. Neurogastroenterol Motil. 2012 Jan;24(1):31-9. doi: 10.1111/j.1365-2982.2011.01803.x. Epub 2011 Nov 9. PMID 22070725
- [Background] Rajilic-Stojanovic M, Heilig HG, Tims S, Zoetendal EG, de Vos WM. Long-term monitoring of the human intestinal microbiota composition. Environ Microbiol. 2012 Oct 15. doi: 10.1111/1462-2920.12023. Online ahead of print. PMID 23286720
- [Background] Simren M, Barbara G, Flint HJ, Spiegel BM, Spiller RC, Vanner S, Verdu EF, Whorwell PJ, Zoetendal EG; Rome Foundation Committee. Intestinal microbiota in functional bowel disorders: a Rome foundation report. Gut. 2013 Jan;62(1):159-76. doi: 10.1136/gutjnl-2012-302167. Epub 2012 Jun 22. PMID 22730468
- [Background] Spiller R, Garsed K. Postinfectious irritable bowel syndrome. Gastroenterology. 2009 May;136(6):1979-88. doi: 10.1053/j.gastro.2009.02.074. Epub 2009 May 7. PMID 19457422
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Yoon JS, Sohn W, Lee OY, Lee SP, Lee KN, Jun DW, Lee HL, Yoon BC, Choi HS, Chung WS, Seo JG. Effect of multispecies probiotics on irritable bowel syndrome: a randomized, double-blind, placebo-controlled trial. J Gastroenterol Hepatol. 2014 Jan;29(1):52-9. doi: 10.1111/jgh.12322. PMID 23829297
- [Background] Youngster I, Russell GH, Pindar C, Ziv-Baran T, Sauk J, Hohmann EL. Oral, capsulized, frozen fecal microbiota transplantation for relapsing Clostridium difficile infection. JAMA. 2014 Nov 5;312(17):1772-8. doi: 10.1001/jama.2014.13875. PMID 25322359
- [Background] Frieling T. [Functional and inflammatory bowel disorders]. Med Klin (Munich). 2006 Mar 22;101 Suppl 1:139-42. German. PMID 16802539
- [Background] Kleger A, Schnell J, Essig A, Wagner M, Bommer M, Seufferlein T, Harter G. Fecal transplant in refractory Clostridium difficile colitis. Dtsch Arztebl Int. 2013 Feb;110(7):108-15. doi: 10.3238/arztebl.2013.0108. Epub 2013 Feb 15. PMID 23468820